CLINICAL TRIAL: NCT06398548
Title: The Impact of 6 Weeks of Moderate- and Heavy-intensity Continous Training on Peak Oxygen Uptake, Plasma Extracellular Vesicles and Inflammatory Cytokines
Brief Title: Impact of Exercise Intensity on Fitness, Extracellular Vesicles, Inflammation, and Metabolism
Acronym: CEX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Jonathan Little, Professor, University of British Columbia
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: H22-02823
Record Dates: First submitted 2024-05-01; First posted 2024-05-03 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Exercise Training
Keywords: Lactate Threshold; Exercise Intensity Domain; VO2peak; Extracellular Vesicles; Mitochondrial Respiration
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: 3 group randomized controlled trial. 1 control group, 2 exercise groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (Other): This group undergoes the same testing protocols as the intervention groups, but is prescribed no additional exercise.
  Interventions: Other: Control Group
- Moderate Intensity Continuous Training (Experimental): In this allocation, participants cycle at 70% the resistance associated with their lactate threshold
  Interventions: Other: Moderate Intensity Continuous Training
- Heavy Intensity Continuous Training (Experimental): In this allocation, participants cycle at the resistance associated with their lactate threshold, with an additional 10% of the difference between their LT and maximal achieved watts during the test.
  Interventions: Other: Heavy Intensity Continuous Training

INTERVENTIONS:
Other: Control Group — Participants continue with their lifestyle as usual, with no modification to lifestyle, or exercise habits.
  Arms: Control Group
Other: Moderate Intensity Continuous Training — This group cycles at 70% of the resistance associated with their first lactate threshold.
  Arms: Moderate Intensity Continuous Training
Other: Heavy Intensity Continuous Training — This group cycles at 10% of the difference between the resistance associated with their lactate threshold, and maximal achieved watts, added to the resistance associated with their lactate threshold.
  Arms: Heavy Intensity Continuous Training

SUMMARY:
Introduction

This study investigates the effects of different intensities of indoor cycling on various health measures. Participants will perform a maximal cycling test to determine their maximal fitness - a strong predictor of overall health - before and after a 6-week training intervention. Blood samples will also be obtained to look at various physiological markers related to extracellular vesicles, inflammation, and metabolism.

Who can participate?

Healthy young adults who between 18 and 40, are free of immune disease, with a normal body mass index can join this study. They will be divided into three groups:

* One group will ride a bike at a moderate pace.
* Another group will ride a bike at a slightly harder pace.
* The third group won't change their usual daily activities and will continue living as they normally do.

What does the study involve?

Each exercise session aims to burn a specific amount of calories: 350 for males and 300 for females. Participants cycle 3 times a week for 6 weeks. At the end, we'll repeat the bike test and take another blood sample to see if there have been any changes due to the exercise.

Why is this research being done?

The researchers want to see how different intensities of exercise impact health and fitness. This may help people make better choices about how much and what type of exercise they should do.

What happens after the study?

Researchers will analyze the data from the study and see if any differences exist between the protocols. If the participant is interested, we will also provide their blood test results, and the results from their max test.

DETAILED DESCRIPTION:
This study is being carried out by the Exercise Metabolism and Inflammation Laboratory at the University of British Columbia campus in Kelowna, British Columbia. Participants who have met the inclusion criteria will first complete an informed consent form. Participants will also complete forms to determine their level of activity. Females will also complete a menstrual cycle questionnaire - but will not be required to start on a particular day in their cycle. Participants will have their anthropometrics recorded (height, weight, body composition), will provide a fasted blood sample, and undergo a maximal staged exercise test to determine their lactate threshold and their maximal oxygen uptake (VO2peak).

The blood test will be used to measure various markers. First, whole blood will be analyzed on a standard hematology analyzer to determine white blood cell counts, red blood cell counts, hemoglobin and platelets. Secondly, blood samples will be spun down to platelet poor plasma and stored for batch analysis. Analysis of plasma will include measurement of plasma cytokines: Interleukin (IL)-6, IL-10, IL-1 receptor agonist, tumor necrosis factor alpha (TNF-alpha) and plasma extracellular vesicles. Extracellular vesicles (EVs) will be isolated using size exclusion chromatography (SEC) and measured for size and concentration using tunable resistive pulse sensing (Izon Exoid, Izon USA). EV phenotype and origin will be determined using nano-flow cytometry (CytoFlex S, Beckman Coulter, USA). EV micro ribonucleic acid (miRNA) will be determined by extracting miRNA from isolated and concentrated EVs (high speed centrifugation of 25,000 x g for 1 hour at 20 degrees Celsius). Extracted miRNA will be measured using PCR (BioRad, USA).

The maximal exercise will occur on a stationary cycle ergometer (Lode Excalibur, Lode, The Netherlands). The ergometer is adjusted to be ideal for each participant. Participants are fitted with a chest strap heart rate monitor (Polar, Finland) and fitted with a face mask to collect to determine the amount of O2 consumption, and CO2¬ production. Lactate measures will be collected from fingertip capillary blood and measured with a lactate analyzer (Nova, USA) during the last 30 seconds of each stage, as is a rating of perceived exertion (RPE). The protocol involves remaining stationary on the ergometer for 2 minutes. Following baseline measures, participants will complete 2 minutes of warm up at 50 watts (W), and then 3-minute stages at consecutively higher workloads (20W increases for females, 30W increases for males). Participants cycle at 60 - 80 revolutions per minute (rpm) for as long as they can. Once they fall below, or cannot maintain a minimum of 50rpm, the test is terminated.

Following the test, the lactate threshold determined as a weighted combination of the log-log method, and Dmax method will be calculated. Weighting consists of 75% of the log-log value and 25% of the Dmax value as calculated in the "lactater" R package. Using their lactate thresholds, specific exercise prescriptions are determined.

Group randomization is completed using a 2:2:1 ratio of moderate intensity continuous training (MICT), heavy intensity continuous training (HICT) and control (CTRL). A power calculation using an alpha of 0.05, power of 0.8 and a medium effect size using changes in VO2peak within the literature suggest that 52 participants will need to complete the study.

For the MICT group, participants will cycle at the resistance associated with 70% of the resistance at their first lactate threshold (LT1) such that if their lactate threshold occurred at 110W, they would initially cycle at 77W (0.7 * 110W). In the HICT group, the participants will cycle at the delta 10% of their lactate threshold and highest achieved resistance at the end of the test. As an example, a participant with a lactate threshold at 110W, who made it to 260W, would cycle at 125W (260W - 110W = 150W), (150W * 0.1 = 15W), (15W + 110W= 125W). Each allocation is matched for energy expenditure, such that males will expend 350 kcals and females will expend 300 kcals.

As the participant progresses through the trial, they will experience an increase in resistance as they adapt to the training protocol. The lactate value associated with their allocation will be maintained throughout. For example, in the 2nd week, if their lactate falls by 10% or more, their resistance will be increased by 10%. The time of each session will also be modified based on the VO2 value associated with their threshold test.

Following the last session of their participation, we will schedule their post test to fall on what would normally be date of their next session. Furthermore, all post testing is completed between 48 and 72 hours following their last session. The post-test and pre-test are identical in nature.

ELIGIBILITY:
Inclusion Criteria:

* Are between the ages of 18 and 40 years old.
* Have a body mass index (BMI) between 18.5 and 30 kg/m^2.
* Perform between 60 and 200 minutes of aerobic physical activity per week.
* Do not have a history of cardiovascular disease or diabetes.

Exclusion Criteria:

* Require immunomodulatory medication to treat an auto-immune disease, or rely heavily on over the counter anti-inflammatory medications (e.g., Advil).
* Have a metabolic condition such as diabetes.
* Have hypertension (blood pressure > 160/90 mmHg).
* Are uncomfortable with blood sampling.
* Are an elite endurance athlete, or training specifically for an endurance event (>3 structured aerobic training sessions, or >150 min of specific aerobic-based/endurance training per week).
* Adhere to an extreme diet (e.g., ketogenic diet, time restricted feeding).
* Smoke cigarettes

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Peak oxygen uptake | 6 Weeks
  The peak oxygen consumption during a maximal staged exercise test

SECONDARY OUTCOMES:
Extracellular Vesicle Phenotype | 6 Weeks
  Plasma extracellular vesicle cellular origin measured by nano-flow cytometry
Extracellular Vesicle Size and Concentration | 6 Weeks
  Plasma extracellular vesicle sizing and concentration measured by tunable resistive pulse sensing.
Extracellular Vesicle micro RNA Content | 6 Weeks
  Plasma extracellular vesicle miRNA content measured by RT-qPCR.
Lactate Threshold | 6 Weeks
  Lactate threshold determined for each participant.
Peak Power Output | 6 Weeks
  Peak power output as measured as the maximal achieved watts during the staged maximal exercise test.
Peripheral Blood Mononuclear Cell Mitochondrial Respiration | 6 Weeks
  Peripheral blood mononuclear cell mitochondrial respiration measured by high resolution respirometry.
Peripheral Blood Mononuclear Cell Gene Expression | 6 Weeks
  The expression of various inflammatory and metabolic genes determined using RT-qPCR

CONTACTS AND LOCATIONS:
Locations (1):
- ART 115, Kelowna, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Yes
De-identified data may be shared based on reasonable request.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data may be available once the manuscript for the study has been published.